CLINICAL TRIAL: NCT05797168
Title: A Modular Phase I/IIa, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Ascending Doses of AZD5335 Monotherapy and in Combination With Anti-cancer Agents in Participants With Solid Tumors
Brief Title: Phase I/IIa Study of AZD5335 as Monotherapy and Combination Therapy in Participants With Solid Tumors
Acronym: FONTANA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8990C00001; 2022-502576-23-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-02-21; First posted 2023-04-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Lung Adenocarcinoma; Endometrial Cancer
Keywords: ADC; PARP inhibitor; AZD5335; AZD5305; Saruparib; Bevacizumab; Carboplatin; AZD9574; Ovarian Cancer; Lung Adenocarcinoma; Endometrial Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Adenocarcinoma of Lung; Endometrial Neoplasms | interventions — AZD5305; Bevacizumab; Carboplatin

STUDY DESIGN:
Intervention Model Description: The study consists of individual modules, each evaluating the safety and tolerability of AZD5335 dosed as monotherapy or in combination with specific treatments.
  * Module 1 (AZD5335 monotherapy)
  * Module 2 (AZD5335 in combination with saruparib)
  * Module 3 (AZD5335 in combination with bevacizumab)
  * Module 4 (AZD5335 in combination with carboplatin +/- bevacizumab)
  * Module 5 (AZD5335 in combination with AZD9574)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Module 1: AZD5335 Monotherapy (Experimental): AZD5335 Monotherapy
  Interventions: Drug: AZD5335
- Module 2: AZD5335 + Saruparib (Experimental): AZD5335 + Saruparib
  Interventions: Drug: AZD5335; Drug: Saruparib (AZD5305)
- Module 3: AZD5335 + Bevacizumab (Experimental): AZD5335 + Bevacizumab
  Interventions: Drug: AZD5335; Drug: Bevacizumab
- Module 4: AZD5335 + Carboplatin +/- Bevacizumab (Experimental): AZD5335 + Carboplatin +/- Bevacizumab
  Interventions: Drug: AZD5335; Drug: Bevacizumab; Drug: Carboplatin
- Module 5: AZD5335 + AZD9574 (Experimental): AZD5335 + AZD9574
  Interventions: Drug: AZD5335; Drug: AZD9574

INTERVENTIONS:
Drug: AZD5335 — IV Antibody-drug conjugate
Drug: Saruparib (AZD5305) — Oral PARP inhibitor
  Other Names: AZD5305
  Arms: Module 2: AZD5335 + Saruparib
Drug: Bevacizumab — IV Monoclonal antibody
  Other Names: Avastin
  Arms: Module 3: AZD5335 + Bevacizumab; Module 4: AZD5335 + Carboplatin +/- Bevacizumab
Drug: Carboplatin — IV Alkylating agent
  Other Names: Paraplatin
  Arms: Module 4: AZD5335 + Carboplatin +/- Bevacizumab
Drug: AZD9574 — Oral PARP inhibitor
  Arms: Module 5: AZD5335 + AZD9574

SUMMARY:
This research is designed to determine if experimental treatment with Antibody-drug conjugate, AZD5335, alone, or in combination with anti-cancer agents is safe, tolerable, and has anti-cancer activity in patients with advanced tumors

DETAILED DESCRIPTION:
This study is a Phase I/IIa modular, open-label, multi-center study of AZD5335 administered either as monotherapy or in combination with other anti-cancer agents in participants with advanced solid malignancies

ELIGIBILITY:
Core Inclusion Criteria:

* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Provision of signed and dated written Optional Genetic Research Information informed consent prior to collection of samples for optional genetic research that supports Genomic Initiative. Participants who do not provide informed consent for Optional Genetic Research may still be enrolled in the study.
* Participant must be ≥ 18 years at the time of signing the informed consent.
* Willing to provide adequate archival and/or baseline tumor sample as applicable per module-specific criteria.
* For participants who have previously received targeted therapies such as ADCs, a fresh baseline biopsy will be required unless the most recent archival tissue sample was collected after receipt of such treatment.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Participants with advanced solid tumors must have received prior adequate therapy in accordance with local practice for their tumor type and stage of disease, or, in the opinion of the Investigator, a clinical trial is the best option for the next treatment based on response and/or tolerability to prior therapy. Participants with contraindications or who refuse therapy in accordance with local practice may also be considered provided that it is documented that he/she was informed about all therapeutic options.
* Participants must have measurable disease per RECIST v1.1,

  1. A previously irradiated lesion can be considered a target lesion if the lesion is progressing and well defined.
  2. For participants who undergo biopsies at screening and/or on treatment, it is preferred though not required, that the biopsied lesion, be distinct from any target lesion used in the RECIST v1.1 evaluation.
* Life expectancy ≥ 12 weeks.
* Adequate organ and marrow function.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  (a) Male participants: (i) Male participants who are sexually active with a female partner of childbearing potential must use a male condom (plus an additional contraceptive method) post-screening through 5 months following the last dose of study intervention. It is strongly recommended for the female partner of a male participant to also use a highly effective method of contraception throughout this period. In addition, male participants must refrain from freezing or donating sperm while on study and for 5 months following the last dose of study intervention.

  (b) Female participants: (i) Females of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study intervention and a negative urine or serum pregnancy test prior to starting their next cycle of treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

(ii) (ii) Sex and Contraceptive/Barrier Requirements: Highly effective birth control methods include: Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the participant (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments) [(periodic abstinence e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to study intervention, and withdrawal are not acceptable methods of contraception], a vasectomized partner, Implanon®, bilateral tubal occlusion, intrauterine device/levonorgestrel intrauterine system, Depo Provera™ injections, oral contraceptive associated with inhibition of ovulation, and Evra Patch™, Xulane™, or NuvaRing®.

Female participants of childbearing potential who are sexually active with a non-sterilized male partner must agree to use one highly effective method of birth control (defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly), from enrolment throughout the study and for 8 months following the last dose of study intervention. The male partner of a female participant of childbearing potential must also use a male condom (plus spermicide, if available) throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. In addition, female participants must not donate or retrieve for their own use, ova while on study and for 8 months following the last dose of study intervention.

Core Exclusion Criteria:

* Patients with spinal cord compression or a history of leptomeningeal carcinomatosis.
* Patients with brain metastases unless, asymptomatic, stable, and not requiring continuous corticosteroids at a dose of > 10 mg prednisone/day or equivalent for at least 4 weeks prior to first dose of study intervention.
* Treatment with any of the protocol defined medications, without adequate washout periods or time before the first dose of study intervention.
* Unresolved toxicities of Grade ≥ 2 (National Cancer Institute [NCI] CTCAE v5.0) from prior therapy (excluding vitiligo, alopecia, and endocrine disorders that are controlled with replacement hormone therapy). Participants with stable ≤ Grade 2 neuropathy are eligible.
* Active infection, including tuberculosis and infections with hepatitis B virus (HBV; verified by known positive hepatitis B surface antigen [HBsAg] result), hepatitis C virus (HCV) or known HIV infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA, CD4+ count ≥ 350/mm3, no history of acquired immune deficiency syndrome-defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on the same anti-HIV medications (meaning there are no expected further changes in that time to the number or type of antiretroviral drugs in the regimen).

Patients with a past or resolved HBV/HCV infection are eligible if:

1. Negative for HBsAg and positive for anti-hepatitis B virus core protein (HBc) or
2. Are HBsAg + with chronic HBV infection (lasting 6 months or longer) and meet conditions i-iii below:

(i) HBV DNA viral load <100 IU/mL. (ii) Have normal transaminase values, or, if liver metastases are present, abnormal transaminases, with a result of aspartate aminotransferase (AST)/alanine aminotransferase (ALT) <3 x upper limit of normal (ULN), which are not attributable to HBV infection.

(iii) Start or maintain antiviral treatment if clinically indicated as per the Investigator or as per local guideline.

Note for Japan: Japanese patients with positive anti-HBs/anti-HBc and negative HBsAg will be assessed following local guidelines.

(c) Participants testing positive for HCV antibody are eligible only if the polymerase chain reaction test result is negative for HCV RNA.

* Patient has ILD/pneumonitis or has a history of (non-infectious) ILD/pneumonitis that required oral or IV steroids or supplemental oxygen, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.

  * Patients with a history of radiation pneumonitis which has clinically and radiologically resolved and not requiring treatment with steroids may be eligible.
* History of another malignancy except for:

  * Malignancy treated with curative intent and with no known active disease for at least 2 years prior to screening of study intervention and with low potential risk for recurrence.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
  * Localized non-invasive solid organ primary disease under surveillance.
* Patients with any of the following cardiac criteria:

  * History of arrhythmia (such as multifocal premature ventricular contractions, bigeminy, trigeminy, and ventricular tachycardia), which is symptomatic or requires treatment NCI CTCAE v5.0 Grade 3 except for:

    (i) Rate controlled asymptomatic atrial fibrillation.
    * NOTE: significant abnormalities in serum electrolytes that can increase the risk of arrhythmic events (ie, sodium, potassium, calcium, and magnesium) should be corrected before starting the study intervention.
  * Uncontrolled hypertension.
  * Acute coronary syndrome/acute myocardial infarction, unstable angina pectoris, coronary intervention procedure with percutaneous coronary intervention, or coronary artery bypass grafting within 6 months of screening.
  * History of brain perfusion problems (eg, carotid stenosis) or stroke, or transient ischemic attack in the last 6 months prior to screening.
  * Symptomatic heart failure (as defined by New York Heart Association class ≥ 2).
  * Prior or current diagnosis of cardiomyopathy considered clinically relevant per investigator's judgement.
  * Severe uncorrected valvular heart disease.
  * Mean resting QTcF > 470 msec obtained from triplicate electrocardiograms (ECGs) and averaged, recorded within 5 minutes.
  * Any factor that, in the opinion of the investigator, increases the proarrhythmic risk of QT prolongation, such as congenital long QT syndrome, family history of long QT syndrome, hypertrophic cardiomyopathy, or unexplained sudden cardiac death under 40 years of age.
* Uncontrolled and/or unresolved intercurrent illness within 12 months prior to screening, including but not limited to serious chronic gastrointestinal conditions associated with diarrhea, or illness (including psychiatric illness) and/or social situations, in the opinion of the investigator, that would limit compliance with study requirements and activities, substantially increase risk of incurring AEs or compromise the ability of the participant to give written informed consent.
* Substance abuse or any other medical conditions that would increase the safety risk to the participant or interfere with participation of the participant or evaluation of the clinical study in the opinion of the Investigator.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention. Note: Participants, if enrolled, should not receive live vaccine whilst receiving study intervention and up to 3 months after the last dose of study intervention. Participants can receive Coronavirus (COVID)-19 vaccines, at the discretion of the Investigator, following a benefit/risk evaluation for the individual participant and in accordance with local rules and regulations and vaccination guidelines. Note: If a COVID-19 vaccine is administered it should be done > 72 hours prior to study intervention initiation or after completion of the DLT period.
* For women only - currently pregnant (confirmed with positive pregnancy test or suspected), lactating, breastfeeding, or intention to become pregnant during the study period.
* Concurrent enrolment in another clinical study, unless it is an observational (non interventional) clinical study or during the follow-up period of an interventional study.
* Patients with a known hypersensitivity to study intervention or any of the excipients of the product.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Previous enrolment in the present study. **Other module specific criteria may apply

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2028-01-06 (Estimated); Study Completion 2028-01-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events/serious adverse events | From time of Informed Consent to 30 days post last dose.
  Number of participants with incidence of adverse events and with serious adverse events including changes from baseline in laboratory parameters, vital signs, ECGs, and physical examination.
The number of participants with dose limiting toxicity(DLT), as defined in the protocol | From the first dose of AZD5335 on Cycle 1 Day 1 up to and including the planned end of Cycle 1 (At the end of 21 days)
  A DLT is defined as any ≥ Grade 3 treatment-emergent AE that occurs during the DLT evaluation period, not attributable to the underlying disease or extraneous causes (as defined in the protocol)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From time of Informed Consent to progressive disease or withdrawal of consent.(approx 2 years)
  The percentage of participants with a confirmed CR or PR according to RECIST v1.1 criteria.
Duration of Response (DoR) | From the first documented response to confirmed progression or death in the absence of disease progression.(approx 2 years)
  The time from the date of first response until date of disease progression or death in the absence of disease progression.
Disease Control Rate (DCR) | From time of Informed Consent until progression.(approx 15 weeks)
  The percentage of participants who have a best objective response of confirmed CR or PR or who have SD for at least 15 weeks after start of treatment (to allow for an early assessment within the assessment window).
Progression free Survival (PFS) | From time of first dose of AZD5335 or AZD5305 until the date of objective disease progression or death (by any cause in the absence of progression).(approx 2 years)
  Progression-free survival is defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the participant withdraws from assigned therapy or receives another anti-cancer therapy prior to progression. Participants who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable RECIST v1.1 assessment
Overall Survival (OS) | From time of first dose of AZD5335 or AZD5305 until death due to any cause.(approx 2 years)
  The time until death due to any cause.
Module 1: Pharmacokinetics of AZD5335: Area Under the concentration-time curve(AUC) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335(approximately 12 weeks)
  Area under the plasma concentration-time curve
Module 1: Pharmacokinetics of AZD5335: Maximum plasma concentration of the study drug (Cmax) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335 (approximately 12 weeks)
  Maximum observed plasma concentration of the study drug
Module 1: Pharmacokinetics of AZD5335: Time to maximum plasma concentration of the study drug (T-max) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335 (approximately 12 weeks)
  Time to maximum observed plasma concentration of the study drug
Module 1: Pharmacokinetics of AZD5335: Clearance | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335 (approximately 12 weeks)
  A pharmacokinetic measurement of the volume of plasma from which the study drug is completely removed per unit time.
Module 1: Pharmacokinetics of AZD5335: Terminal elimination half-life (t 1/2) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335 (approximately 12 weeks)
  Terminal elimination half life.
Immunogenicity of AZD5335 | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5535.(approx 2 years)
  The number and percentage of participants who develop ADAs.
Module 1: To investigate baseline and on treatment changes in target expression. | Baseline and predicted intervals throughout the administration of AZD5335(approx 2 years)
  The clinical activity by baseline and on-treatment changes in tumor target expression.
Module 2: Pharmacokinetics of AZD5335 and AZD5305 when given in combination. | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335 and AZD5305.(approx 12 weeks)
  The plasma concentrations of AZD5335, total antibody, and total unconjugated payload.
Module 2, 3, 4, and 5: Area Under the concentration-time curve (AUC) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  Area under the plasma concentration-time curve
Module 2, 3, 4, and 5: Maximum plasma concentration of the study drug (Cmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  Maximum observed plasma concentration of the study drug
Module 2, 3, 4, and 5: Time to maximum plasma concentration of the study drug (T-max) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  Time to maximum observed plasma concentration of the study drug
Module 2, 3, 4, and 5: Clearance | At predefined intervals throughout the treatment period (approximately 12 weeks)
  A pharmacokinetic measurement of the volume of plasma from which the study drug is completely removed per unit time.
Module 2, 3, 4, and 5: Terminal elimination half-life (t 1/2) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335 (approximately 12 weeks)
  Terminal elimination half life.
Module 3: Pharmacokinetics of AZD5335 and bevaczizumab when given in combination. | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335 and bevacizumab.(approx 12 weeks)
  The plasma concentrations of AZD5335, total antibody, and total unconjugated payload.
Module 4: Pharmacokinetics of AZD5335 and carboplatin (+/- bevacizumab) when given in combination. | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335 and carboplatin (+/- bevacizumab).(approx 12 weeks)
  The plasma concentrations of AZD5335, total antibody, and total unconjugated payload.
Module 5: Pharmacokinetics of AZD5335 and AZD9574 when given in combination. | From the first dose of study intervention, at predefined intervals throughout the administration of AZD5335 and AZD9574.(approx 12 weeks)
  The plasma concentrations of AZD5335, total antibody, and total unconjugated payload.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (51):
- United States (12):
  - Research Site, Duarte, California
  - Research Site, Irvine, California
  - Research Site, La Jolla, California
  - Research Site, Aurora, Colorado
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Providence, Rhode Island
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Australia (2):
  - Research Site, Liverpool
  - Research Site, Melbourne
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (6):
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Jinan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Germany (7):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Mannheim
  - Research Site, Regensburg
- Israel (2):
  - Research Site, Haifa
  - Research Site, Ramat Gan
- Japan (5):
  - Research Site, Hidaka-shi
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Sunto-gun
  - Research Site, Tokyo
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Istanbul
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Glasgow, Scotland
  - Research Site, London
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home